CLINICAL TRIAL: NCT02708004
Title: A Single-center, Double-blind, Randomized, Placebo-controlled, Two-way Crossover Study to Assess Body Fluid Homeostasis After Administration of ACT-132577 in Healthy Subjects
Brief Title: Clinical Study to Assess Body Fluid Homeostasis After Administration of ACT-132577 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AC-080-102
Record Dates: First submitted 2016-02-24; First posted 2016-03-15 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — aprocitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT-132577 (Experimental): 3 different dose levels
  Interventions: Drug: Aprocitentan
- Placebo (Placebo Comparator): Matching active drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aprocitentan — Formulated in capsules in 2 different strengths; 2 capsules per day
  Other Names: ACT-132577
  Arms: ACT-132577
Other: Placebo — Matching active drug
  Arms: Placebo

SUMMARY:
This clinical study will be conducted to evaluate the effect of ACT-132577 on fluid homeostasis in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy on the basis of medical history, physical examination, cardiovascular assessments and hematology, clinical chemistry, and urinalysis tests
* Body mass index between 20.0 and 25.0 kg/m2 (inclusive) at screening

Exclusion Criteria:

- Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-01; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Body weight | from Day 1 to Day 9
  Change from baseline

OTHER OUTCOMES:
Treatment-emergent Adverse Events | From Day 1 up to End-of-Study (i.e. for at least 25 days)
  Number of subjects with Adverse Events
Treatment-emergent Serious Adverse Events | From Screening (Day -3) up to Follow-up (i.e. for at least 49 days)
  Number of subjects with Serious Adverse Events
Glomerular filtration rate (GFR) | At 0 h of Day 1, at 1 h, 2 h, 4 h, 6 h and 10 h of Day 1 & Day 9
  Change from baseline to each scheduled timepoint
Fractional sodium excretion in 24 h urine samples [mmol per day] | At 0 h of Day 1, at 1 h, 2 h, 4 h, 6 h and 10 h of Day 1 & Day 9
  Fractional excretion will be calculated as the clearance of sodium divided by the clearance of creatinine. Change from baseline to each scheduled timepoint
Fractional lithium excretion in 24 h urine samples [mmol per day] | At 0 h of Day 1, at 1 h, 2 h, 4 h, 6 h and 10 h of Day 1 & Day 9
  Fractional excretion will be calculated as the clearance of lithium divided by the clearance of creatinine. Change from baseline to each scheduled timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Investigator Site Lausanne, Lausanne, Switzerland